CLINICAL TRIAL: NCT05781126
Title: The Effect of Listening Effort, Cognition Status, and Anxiety or Depression in Listening Satisfaction by Hearing Aid Users
Brief Title: The Effect of Listening Effort, Cognition and Anxiety-depression in Listening Satisfaction by Hearing Aid Users
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chania General Hospital "St. George" (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Sponsor
Other Study IDs: ENT_CHANIA_02
Record Dates: First submitted 2023-01-23; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-01

CONDITIONS: Listening Effort; Cognitive Function 1, Social; Anxiety; Depression; Satisfaction, Consumer; Amplification; Hearing Aid
MeSH Terms: conditions — Anxiety Disorders; Depression; Consumer Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: The Spatial Hearing Questionnaire, MINI-MENTAL STATE EXAMINATION, International Outcome Inventory - Hearing Aid, Glasgow Hearing Aid Benefit Profile, BECK-II and STAI questionnaires — a) medical history record, b) ENT examination, c) pure tone audiogram and speech audiometry (with and without the hearing amplification) d) listening effort evaluation (with and without the hearing amplification) Self-report and behavioral methods will be used: Evaluation of subjective performance (Spatial Hearing Questionnaire (SHQ) Evaluation of time response in auditory message Evaluation of speech comprehension with background noise or a competitive speaker e) cognitive function evaluation by using the Greek version of Mini-Mental State Examination, f) evaluation of hearing-aid satisfaction, by using the Glasgow Hearing Aid Benefit Profile (GHABP), and International Outcome Inventory - Hearing Aid (IOI-HA), questionnaires and g) evaluation of stress level and depression by using BECK-II and STAI questionnaires.

SUMMARY:
Brief Summary Introduction: Listening can be effortful in situations that require the intensive use of cognitive processing resources especially for individuals with a hearing loss. Hearing-impaired listeners are under a greater degree of cognitive challenge during a hearing task, speech comprehension, memory, response in an auditory message. Listening effort is defined as 'the attention and cognitive resources required to understand speech'. Hearing ability is the strongest predictor of speech understanding accuracy, but cognitive factors, psychological state of the listener and stress also play a significant role. Although there is no gold-standard method for listening effort assessment. a wide range of techniques is used such as: a) self-report methods, b) behavioral measures, or c) physiological measures. Cognitive functioning refers to multiple mental abilities, including receiving visual and auditory message, decision making, processing information and memory skills. During the ageing process there is a decline in cognitive function. The most common tools to measure it are: a) Montreal Cognitive Assessment (MoCA) test b) Mini-Mental State Exam (MMSE), and c) το Mini Cog. Within the older adult population with hearing loss, prevalence estimates that up to 20% report a clinically relevant level of depression symptoms that would necessitate treatment. A cross-sectional association between hearing loss and depression among older adults has been consistently observed. A reduction in activities of daily living observed in older adults with hearing loss, suggesting that disengagement in activities post-hearing loss may contribute to depression. The satisfaction due to amplification for the hearing aid- user is effected by the changes in his everyday routine and also depend on the level of his cognitive function, motivation, psychological status and social environment. Purpose: The purpose of this study is to investigate the effect of listening effort, cognitive function, stress and depression on amplification satisfaction for adult hearing aid-users. Methods and materials: This is a prospective study including patients examined in the outpatient department of ENT clinic in General Hospital of Chania. Patients fulfilling the inclusion criteria will undergo: a) medical history record, b) ENT examination, c) pure tone audiogram and speech audiometry (with and without the hearing amplification) d) listening effort evaluation (with and without the hearing amplification) Self-report and behavioral methods will be used: Evaluation of subjective performance (Spatial Hearing Questionnaire (SHQ) Evaluation of time response in auditory message Evaluation of speech comprehension with background noise or a competitive speaker e) cognitive function evaluation by using the Greek version of Mini-Mental State Examination, f) evaluation of hearing-aid satisfaction, by using the Glasgow Hearing Aid Benefit Profile (GHABP), and International Outcome Inventory - Hearing Aid (IOI-HA), questionnaires and g) evaluation of stress level and depression by using BECK-II and STAI questionnaires. Results: The main outcome will be the assessment of listening effort, cognitive function, psychological status (stress/depression) effect on the level of satisfaction of hearing-aid users. Additional outcomes will be the assessment of the effect of cognitive decline in listening effort and the effect of psychological status on listening effort. Study findings will highlight the potential of changing the approach and management of the hearing aid-users in a way that hearing amplification will lead to satisfaction of their expectations

ELIGIBILITY:
Inclusion Criteria:

1. participants aged between 18 and 80 years
2. with sensorineural or mixed bilateral hearing loss
3. wearing a hearing aid, unilaterally or bilaterally for at least 6 months
4. all participants should give a written consent for their participation and the permission for the anonymously use of their results.

Exclusion Criteria:

1. known neurological disease e.g. neurodegenerative disease (including disease Alzheimer's or dementia), demyelinating disease, metastatic disease
2. known psychiatric illness
3. illiteracy or non-use of the Greek language
4. non-consent to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the outpatient ENT clinic of Chania General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Hearing aid users satisfaction | 20 minutes
  Glasgow Hearing Aid Benefit Profile (GHABP), patients choose and answer from 0-5 where 0 is the worst result and 5 the best about their satisfaction
  International Outcome Inventory - Hearing Aid (IOI-HA) patients choose one answer between five beginning from the worst feeling to the best (not helping/not worth it/worse - moderate - very helpful/totally worth it)
Listening effort | 40 minutes
  Spatial Hearing Questionnaire (SHQ), in which patients rate from 0-100 each question (0 is the worst condition and 100 the best)
  Intelligibility test in noise Time response in intelligibility test
Cognitive function | 15 minutes
  Mini-Mental State Examination, 1 point for each correct answer maximun score: 30 - minimum score:24
Anxiety or depression | 20 minutes
  State-Trait Anxiety Inventory (STAI) .Higher scores are positively correlated with higher levels of anxiety
  Beck's Depression Inventory (BECK-II) Higher total scores indicate more severe depression
Listening effort and cognitive impairment. | 10 minutes
  Correlation between intelligibility test results, and time response, Spatial Hearing Questionnaire (SHQ) and Mini-Mental State Examination
Listening effort and Hearing aid users satisfaction | 10 minutes
  Correlation between intelligibility test results, and time response, Spatial Hearing Questionnaire (SHQ) and Glasgow Hearing Aid Benefit Profile (GHABP), International Outcome Inventory - Hearing Aid (IOI-HA)
Hearing aid users satisfaction and Anxiety or depression | 10 minutes
  Correlation between Glasgow Hearing Aid Benefit Profile (GHABP), International Outcome Inventory - Hearing Aid (IOI-HA) and State-Trait Anxiety Inventory (STAI), Beck's Depression Inventory (BECK-II)
Listening effort and Anxiety or depression | 10 minutes
  Correlation between intelligibility test results, and time response, Spatial Hearing Questionnaire (SHQ) and State-Trait Anxiety Inventory (STAI), Beck's Depression Inventory (BECK-II)

CONTACTS AND LOCATIONS:
Overall Officials: Chariton Papadakis, MD, PhD, Study Chair — Chania General Hospital "St. George"